CLINICAL TRIAL: NCT00954070
Title: Detection of Minimal Change Esophagitis Using Confocal Laser Endomicroscopy
Status: Terminated | Type: Observational
Why Stopped: Difficulty in recruiting subjects for study
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Medicine, Professor & Senior Consultant Gastroenterologist, National University Hospital, Singapore
Other Study IDs: E/09/026
Record Dates: First submitted 2009-07-08; First posted 2009-08-06 (Estimated); Last update posted 2012-12-28 (Estimated); Status verified 2012-12

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: gastroesophageal reflux disease
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case (subjects with NERD): The investigators cases are subjects with confirmed NERD and include male or female patients aged between 21 and 65 years, who present with typical clinical manifestations of gastroesophageal reflux and have no esophageal mucosal breaks upon conventional white-light endoscopy examination but show evidence of pathologic gastroesophageal reflux on 24-hr pH monitoring.
  Interventions: Device: Confocal endomicroscope (Pentax Model EC3870K)
- Control: Healthy individuals aged between 21 and 65 years who are asymptomatic for GERD and other digestive diseases
  Interventions: Device: Confocal endomicroscope (Pentax Model EC3870K)

INTERVENTIONS:
Device: Confocal endomicroscope (Pentax Model EC3870K) — The intervention is an endoscopy procedure using a novel type of endoscope with a powerful confocal microscope attached to its tip. The endoscope (Pentax Model EC3870K) provides both white-light and confocal microscopic imaging.
  Other Names: Pentax Model EC3870K, Pentax Corp, Tokyo, Japan

SUMMARY:
This is an observational, prospective and pilot study to determine through confocal endomicroscopy diagnostic microscopic features detectable at the gastroesophageal junction of patients with non-erosive gastroesophageal reflux disease.

The hypothesis is that minimal mucosal changes occur in non-erosive gastroesophageal reflux disease. Although these minimal changes are not always visible on white-light endoscopy, it is detectable using high-resolution confocal endomicroscopy and these confocal features are diagnostic of non-erosive reflux disease (NERD).

DETAILED DESCRIPTION:
In Asia, up to 70% of patients with typical gastroesophageal reflux symptoms could have non-erosive reflux disease (NERD), in which case, no detectable mucosal break may be observed on conventional white-light endoscopy. However, minimal change lesions are often visible upon high-resolution endoscopy and on microscopic examination of biopsied specimens. The most commonly seen microscopic features are dilated intercellular space, infiltration of inflammatory cells into squamous epithelia, hyperplasia of the epithelial basal cell and elongation of the papillae. So far, the most consistent histologic change found in NERD has been the dilated intercellular space in esophageal epithelium. But until now, determinations of intercellular space dilatations could only be done ex-vivo on biopsy specimens using transmission electron microscopy or light microscopy. With the advent of high-resolution confocal laser endomicroscopy, in-vivo determination of intercellular space dilatations and other diagnostic microscopic features could be a reality. This study is aimed at exploring such a clinical possibility and feasibility, with the intention of comparing the microscopic findings based on confocal endomicroscopy with that of symptoms, and esophageal pH.

ELIGIBILITY:
Inclusion Criteria:

* Cases:

  * male or female patients aged between 21 and 65 years with typical clinical manifestations of gastroesophageal reflux but endoscopy-negative for esophageal mucosal breaks
  * by typical clinical manifestations of gastroesophageal reflux, we refer to the occurrence of heartburn and/or regurgitation more than twice a week, with a minimum duration of 8 consecutive weeks, and with symptoms severe enough to affect daily activities
* Controls:

  * healthy male or female aged between 21 and 65 years who are asymptomatic for GERD and other digestive diseases

Exclusion Criteria:

* Endoscopic confirmed erosive esophagitis
* Complications such as Barrett's esophagus, gastric and/or duodenal peptic ulcer, stenosis
* Esophageal, gastric or duodenal cancer or other malignancy
* History of esophagus, stomach, or duodenum surgery
* Conditions that preclude safe biopsies (coagulopathy, haemophilia, esophageal varices, and patients on warfarin and antiplatelets)
* Scleroderma, diabetes mellitus, autonomic or peripheral neuropathy, myopathy or any underlying disease or medication that might affect the lower esophageal sphincter pressure or increase the acid clearance time
* A history of bronchial asthma, or known allergy to fluorescein
* Pregnant or breast-feeding (for females)
* Below 21 or above 65 years of age
* Severe co-morbidities (e.g., such as end-stage renal failure, congestive cardiac failure, liver cirrhosis, severe arthritis requiring long term non-steroidal anti-inflammatory drug therapy)
* Unable or unwilling to give informed consent

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hosipital patients with typical clinical manifestations of gastroesophageal reflux disease but no endoscopy evidence of esophagitis.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2009-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Specific microscopic changes in the esophageal mucosa as seen under the confocal endomicroscope | After 4 weeks phamacological washout period

CONTACTS AND LOCATIONS:
Overall Officials: Khek Yu Ho, MD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Barlow WJ, Orlando RC. The pathogenesis of heartburn in nonerosive reflux disease: a unifying hypothesis. Gastroenterology. 2005 Mar;128(3):771-8. doi: 10.1053/j.gastro.2004.08.014. PMID 15765412
- [Background] Calabrese C, Fabbri A, Bortolotti M, Cenacchi G, Areni A, Scialpi C, Miglioli M, Di Febo G. Dilated intercellular spaces as a marker of oesophageal damage: comparative results in gastro-oesophageal reflux disease with or without bile reflux. Aliment Pharmacol Ther. 2003 Sep 1;18(5):525-32. doi: 10.1046/j.1365-2036.2003.01713.x. PMID 12950425
- [Background] Ravelli AM, Villanacci V, Ruzzenenti N, Grigolato P, Tobanelli P, Klersy C, Rindi G. Dilated intercellular spaces: a major morphological feature of esophagitis. J Pediatr Gastroenterol Nutr. 2006 May;42(5):510-5. doi: 10.1097/01.mpg.0000215312.78664.b9. PMID 16707972
- [Background] Caviglia R, Ribolsi M, Gentile M, Rabitti C, Emerenziani S, Guarino MP, Petitti T, Cicala M. Dilated intercellular spaces and acid reflux at the distal and proximal oesophagus in patients with non-erosive gastro-oesophageal reflux disease. Aliment Pharmacol Ther. 2007 Mar 1;25(5):629-36. doi: 10.1111/j.1365-2036.2006.03237.x. PMID 17305764
- [Background] Caviglia R, Ribolsi M, Maggiano N, Gabbrielli AM, Emerenziani S, Guarino MP, Carotti S, Habib FI, Rabitti C, Cicala M. Dilated intercellular spaces of esophageal epithelium in nonerosive reflux disease patients with physiological esophageal acid exposure. Am J Gastroenterol. 2005 Mar;100(3):543-8. doi: 10.1111/j.1572-0241.2005.40978.x. PMID 15743349